CLINICAL TRIAL: NCT01626105
Title: Study of Severe Hemophilia A Patients Who Have Only Received a Single Recombinant FVIII Therapeutic for the Purpose of Identifying the Pharmacogenetic Determinants of Tolerance and Immunogenicity
Brief Title: Personalized Prediction of Tolerance and Immunogenicity in Hemophilia
Acronym: PPTIH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Victor J Marder, M.D. (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor-Investigator, Victor J Marder, M.D., Associate Professor, Director Hemostasis, Pathology, Veterans Affairs Greater Los Angeles, Los Angeles Orthopaedic Hospital
Organization: Los Angeles Orthopaedic Hospital (Other)
Other Study IDs: PPTIH No. 1
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; Factor VIII; Inhibitors; Immunogenicity; Pharmacogenetics; Mutation; Nonsynonymous Single Nucleotide Polymorphisms; Class II Human Leukocyte Antigens
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A core laboratory exists for this study and will house a Biorepository containing the following:
  1. White blood cells
  2. Blood plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is designed to accurately identify the pharmacogenetic determinants of risk of Factor VIII (FVIII) inhibitor development by focusing on only a select group of Hemophilia A (HA) patients who have: (i) received a recombinant FVIII therapeutic product containing the same primary amino acid sequence since their original diagnosis; (ii) verifiable FVIII infusion histories; and (iii) been tested regularly for FVIII inhibitor development.

DETAILED DESCRIPTION:
We are developing a novel, personalized strategy for assessing immunogenicity of protein therapeutics using, as our model, the infusion of Factor VIII (FVIII) into hemophilia A (HA) patients. About 20% of all treated HA patients develop neutralizing FVIII alloantibodies ("inhibitors") that make disease management difficult and expensive. Nowadays, HA is usually treated with highly purified human recombinant (r)-proteins, an advance in safety from pathogens not accompanied by a decrease in inhibitor incidence. Current strategies for upcoming FVIII formulations focus largely on engineering the most immunogenic epitopes in the hope of forming a universally less immunogenic protein. In contrast, we are pioneering a pharmacogenetic approach to immunogenicity that takes into account the underlying variability of the patient population.

This project focuses on defining the role of individual genetic differences on FVIII immunogenicity. The principles, however, have broader application for protein therapeutics in general. We have studied non-HA-causing variants in the FVIII gene (F8) and have shown that (i) nonsynonymous (ns)-single-nucleotide polymorphisms (SNPs) encode several structurally distinct wild-type FVIII proteins in the human population and (ii) a sequence mismatch between patients' endogenous FVIII and infused FVIII due to ns-SNPs is a risk factor for inhibitor development that may explain the high inhibitor incidence in HA patients with black African ancestry.

The most well established risk factor for inhibitor development is the type of HA-causing F8 gene mutation. As a rule, large alterations in F8 and absence of antigenically cross-reactive material (CRM) in plasma are associated with inhibitor development. The most common F8 mutation causing severe HA, an intron-22-inversion (I22I), fits that description but is not associated with a high inhibitor risk. Similarly, while most HA patients with missense mutations do not develop inhibitors, this alloimmune complication occurs frequently in patients with one of a few highly recurrent missense mutations.

While not definitively established, population heterogeneity in the repertoires of HLA-class-II (HLA-II) molecules expressed on the surfaces of the antigen-presenting cells in individual patients is likely another genetic contributor to inhibitor risk.

This project is a comprehensive assessment of the pharmacogenetics of the immune response to FVIII leveraging a unique resource comprised of a group of 55 subjects with severe or moderately-severe HA who were (i) enrolled as previously-untreated patients (PUPs) in the recently concluded clinical trial known as the Advate PUP study and (ii) have received the same r-FVIII protein (i.e., Advate) since birth. Prior PUP-study data as well as new blood samples and data will be obtained from these subjects upon their enrollment into the current study. In addition to having been treated with only a single FVIII product, this exceptional patient cohort was (and continues to be) closely monitored for both FVIII infusion history and inhibitor development, the latter of which by undergoing frequent Bethesda testing. (HA patients who have been treated with several FVIII products are not ideal for testing the hypotheses we have proposed.)

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe or moderately severe hemophilia A (HA) who have since birth been treated with only a single Factor VIII product (i.e., FVIII protein molecules containing only one primary amino acid sequence).

Exclusion Criteria:

* HA patients with severities other than severe or moderately severe.
* Hemophilia B patients.
* HA patients who have been treated with more than one FVIII product.
* HA patients who have been treated with more than one FVIII product.
* HA patients who do not have verifiable infusion histories.
* HA patients who lack documentable inhibitor testing & infusion histories.

Min Age: 2 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Fifty five patients with severe or moderately severe hemophilia A who have received replacement therapy with a Factor VIII product representing only a single primary amino acid sequence.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-04 (Estimated); Study Completion 2014-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Victor J. Marder, M.D., Principal Investigator — The Los Angeles Orthopaedic Hospital and The David Geffen School of Medicine at UCLA
Locations (1):
- Children's Hospital of Michigan, Detroit, Michigan, United States

REFERENCES:
- [Background] Yanover C, Jain N, Pierce G, Howard TE, Sauna ZE. Pharmacogenetics and the immunogenicity of protein therapeutics. Nat Biotechnol. 2011 Oct 13;29(10):870-3. doi: 10.1038/nbt.2002. No abstract available. PMID 21997623
- [Background] Howard TE, Yanover C, Mahlangu J, Krause A, Viel KR, Kasper CK, Pratt KP. Haemophilia management: time to get personal? Haemophilia. 2011 Sep;17(5):721-8. doi: 10.1111/j.1365-2516.2011.02517.x. Epub 2011 Jun 8. PMID 21649795
- [Background] Viel KR, Ameri A, Abshire TC, Iyer RV, Watts RG, Lutcher C, Channell C, Cole SA, Fernstrom KM, Nakaya S, Kasper CK, Thompson AR, Almasy L, Howard TE. Inhibitors of factor VIII in black patients with hemophilia. N Engl J Med. 2009 Apr 16;360(16):1618-27. doi: 10.1056/NEJMoa075760. PMID 19369668
- See also: The Keck School of Medicine of USC — http://keck.usc.edu/
- See also: The Los Angeles Orthopaedic Hospital in Alliance with UCLA Health System — http://www.orthohospital.org/